CLINICAL TRIAL: NCT05760183
Title: An Observational Medical Trial Assessing Patterns in Experiences of Participants of Metastatic Breast Cancer Clinical Trials
Brief Title: Discovering Factors in Metastatic Breast Cancer Patients' Clinical Trial Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82944089
Record Dates: First submitted 2023-02-25; First posted 2023-03-08 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Enrollment in clinical trials usually favors a particular demographic group. But there is limited research available to explain what study attributes affect the completion of these specific demographic groups.

This trial will evaluate the safety and efficacy of metastatic breast cancer treatments. The focus will be on tracking the rates of completion and withdrawal among these individuals.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future metastatic breast cancer studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient is able and willing to comply with the treatment/follow-up schedule and requirements
* Patient must provide written informed consent

Exclusion Criteria:

* Women who are pregnant, intend to become pregnant, or are lactating
* Inability to perform regular electronic reporting
* Participants who are vulnerable to any intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are actively considering involvement in an observational metastatic breast cancer clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a metastatic breast cancer clinical study. | 3 months
Number of metastatic breast cancer study participants who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conde-Estevez D, Tusquets I, Servitja S, Martinez-Garcia M, Salas E, Albanell J. An overview of randomized clinical trials in metastatic breast cancer: variables affecting regulatory drug approval. Anticancer Drugs. 2014 Oct;25(9):992-7. doi: 10.1097/CAD.0000000000000130. PMID 24892723
- [Background] Kuerer HM, van la Parra RF. Breast Cancer Clinical Trials: Past Half Century Moving Forward Advancing Patient Outcomes. Ann Surg Oncol. 2016 Oct;23(10):3145-52. doi: 10.1245/s10434-016-5326-9. Epub 2016 Jun 30. PMID 27364503
- [Background] Ghislain I, Zikos E, Coens C, Quinten C, Balta V, Tryfonidis K, Piccart M, Zardavas D, Nagele E, Bjelic-Radisic V, Cardoso F, Sprangers MAG, Velikova G, Bottomley A; European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Group; Breast Cancer Group; EORTC Headquarters. Health-related quality of life in locally advanced and metastatic breast cancer: methodological and clinical issues in randomised controlled trials. Lancet Oncol. 2016 Jul;17(7):e294-e304. doi: 10.1016/S1470-2045(16)30099-7. PMID 27396647

DOCUMENTS (1):
  • Informed Consent Form (2023-02-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT05760183/ICF_000.pdf